CLINICAL TRIAL: NCT05112796
Title: Vestibular Socket Therapy (VST) Versus Partial Extraction Therapy (PET) for Treating Fresh Extraction Sites With Thin Labial Plate of Bone With Immediate Implant Placement in the Esthetic Zone: A Randomized Clinical Trial
Brief Title: Vestibular Socket Therapy (VST) Versus Partial Extraction Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VST_PET_20
Record Dates: First submitted 2021-10-29; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Dental Implants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VST technique (Experimental)
  Interventions: Procedure: Class I extractions sites received immediate implants using the Vestibular Socket Therapy
- PET technique (Active Comparator)
  Interventions: Procedure: class I extractions sites received immediate implants using the Partial Extraction Therapy

INTERVENTIONS:
Procedure: Class I extractions sites received immediate implants using the Vestibular Socket Therapy — A 1-cm-long vestibular access incision was made using a 15c blade 3 to 4 mm apical to the mucogingival junction at the related socket. A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision
  Arms: VST technique
Procedure: class I extractions sites received immediate implants using the Partial Extraction Therapy — the hopeless tooth was decoronated 1 mm coronal to the gingival margin using a diamond bur. Then, the facial root segment was separated from the rest of the root using a Lindemann bur in gentle mesiodistal sweeping strokes from the gingival margin to the apex of the root, aiming to separate the palatal and the labial root segments.
  Arms: PET technique

SUMMARY:
The current randomized clinical trial aimed to compare the VST versus Partial Extraction Therapy (PET) for immediate implant placement in the esthetic zone in class I fresh extraction sites.

The primary outcome was the assessment of vertical dimensional changes in peri-implant soft tissue margin.

The secondary outcome was the assessment of radiographic changes in the thickness of the facial peri-implant tissues.

ELIGIBILITY:
Inclusion Criteria:

* single hopeless maxillary tooth in the esthetic zone
* non-smokers
* systemically healthy
* Class I extraction sites

Exclusion Criteria:

* smoking
* Class II and III extraction sites
* hopeless teeth with acute infection or vertical/horizontal root fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Changes in the peri-implant facial tissue thickness | at baseline and 6 months
  through CBCT images (Carestream 8000D- Carestream Dental) that were taken at baseline and 6 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Private Practice Clinic, Alexandria, Egypt